CLINICAL TRIAL: NCT03071250
Title: An Analysis of the Outcomes From Protocolized Perioperative Care for Patients Receiving Total Hip or Knee Arthroplasty
Status: Completed | Type: Observational
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Other Study IDs: 206501
Record Dates: First submitted 2017-03-01; First posted 2017-03-06 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Knee Osteoarthritis; Hip Osteoarthritis; Knee Arthritis; Hip Arthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis, Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Total knee or Hip Arthroplasty — Patients who received either a total knee or hip arthroplasty will be identified

SUMMARY:
The care for patients receiving total hip and knee arthroplasty at the University of Arkansas for Medical Sciences has followed a structured care pathway since July 2015. This system of perioperative care has focused on preoperative assessment of medical co-morbidities and risks to postoperative functional recovery, anesthetic care focused on postoperative nausea and vomiting prevention and optimizing immediate postoperative functional ability, and aggressive postoperative physical therapy.

This is an observational study to look at the outcomes of this program at University of Arkansas for Medical Sciences. Areas of focus will be hospital length of stay, postoperative narcotic consumption, Visual Analog Scale scores, incidence of postoperative nausea and vomiting, and 30-day readmission rates, and health literacy rates.

ELIGIBILITY:
Inclusion Criteria:

- All men and women 18 years and older who underwent total hip arthroplasty or total knee arthroplasty surgery at UAMS between 7/01/2015 and 7/01/2016.

Exclusion Criteria:

- none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects must meet all of the inclusion and exclusion criteria to be enrolled in the study.
  All men and women 18 years and older who underwent total hip arthroplasty or total knee arthroplasty surgery at UAMS between 7/01/2015 and 7/01/2016.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Length of Stay | 7/1/2015 - 7/1/2016
  Postoperative hospital length of stay

SECONDARY OUTCOMES:
narcotic consumption | 7/1/2015 - 7/1/2016
  30-day postoperative narcotic consumption
Pain scores | 7/1/2015 - 7/1/2016
  postoperative VAS pain scores
30-day readmission | 7/1/2015 - 7/1/2016
  30-day hospital readmission following procedure
infection | 7/1/2015 - 7/1/2016
  Surgical site infections
PONV | 7/1/2015 - 7/1/2016
  postoperative nausea and vomiting

CONTACTS AND LOCATIONS:
Locations (1):
- University of Arkansas for MEdical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No